CLINICAL TRIAL: NCT05013528
Title: Comparative Effect of Rhythmic Balance Auditory Vision Training (Bal-A-Vis-X) and Aerobic Training in Children With Autism Spectrum Disorder
Brief Title: Balance Auditory Vision Training (Bal-A-Vis-X) and Aerobic Training in Children With Autism Spectrum Disorder
Acronym: Bal-A-Vis-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00826 Mahnoor Zia
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Aerobic Training; Autism Spectrum Disorder; Bal-A-Vis-X; Balance Auditory Vision Training
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither subjects nor the investigator who is assessing the patient are aware of the treatment assignment until the end of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bal-A-Vis-X training Group (Experimental): Bal-A-Vis-X training Group
  Interventions: Other: Bal-A-Vis-X training; Other: Aerobic Training Group
- Aerobic Training Group (Active Comparator): Aerobic Training Group
  Interventions: Other: Bal-A-Vis-X training; Other: Aerobic Training Group

INTERVENTIONS:
Other: Bal-A-Vis-X training — Bal-A-Vis-X training Performed thrice a week for 10 minutes after baseline assessment Standard Physical therapy treatment along with following exercises.
  1. ball Rectangle
  2. ball rectangle and 2 ball drop/pass/catch two-foot jumping forward, tandem walking on ground and tandem walking on the balance beam. .
  Other Names: Group A
Other: Aerobic Training Group — Aerobic training group performed exercises thrice a week for 10 minutes after baseline assessment.
  Standard Physical therapy treatment along with aerobic training as Running is performed
  Other Names: Group B

SUMMARY:
the aim of this study is to compare the effects of Rhythmic Balance, Auditory, and Vision Exercises and Aerobic training in children with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
Autism is an Umbrella term for a lifelong neuropsychiatric disorder which falls into the category of pervasive developmental disabilities. Autistic Spectrum Disorder (ASD) is a syndrome that often develops in early childhood, characterized by impairment of speech, the problems encountered in communication with the environment, display of certain skills, and developmental retardation in almost all cognitive functions. Autism is a "spectrum disorder'' ranging in severity in every individual. Symptoms of autistic disorder arise during the initial 2 years of life. Problem with language advancement and social interaction are the major concerns reported by parents by 2 years of age.

Evidence has recommended that motor disability is quite possibly the most predictable markers, close by socio communicative challenges, for mental imbalance range issue such as autism spectrum disorder. These motor anomalies could have basic ramifications for resulting psychological and social turn of events. In any case, this territory of improvement is especially under examined in the mental imbalance related setting, and early mediation programs normally center around the core symptoms of the Autism disorder. Although the confined nature of the literature prevents researchers from drawing definitive conclusions, the outcomes from the research mentioned in this study verified probably huge upgrades in the motor skills of autistic children after the physical therapy interventions.

Physical activity plays important role in improving cognition, enhancing executive functions of children to perform daily life activities in children with Autism Spectrum disorders and mental retardation A case report organized and ratified by Rehabilitation department of the University of Lowa, to determine the efficacy of Rhythmic Balance, Auditory, and Vision Exercises as an adjunctive intervention to conventional physical therapy protocol administered in child with Autism and ADHD.A 6 year old child diagnosed with ADHD and Autism was recruited in the study with major recognized difficulties in strength and agility. A 9 week protocol of Bal-A-Vis-X program involving a multi system approach was incorporated in addition to basic pediatric rehabilitation protocol. A notable improvement in child gross motor functions was observed as measured by Bruininks-Oseretsky Test of Motor Proficiency, Second Edition after the intervention.

A pilot study was conducted to ascertain the effect of Rhythmic Balance, Auditory, and Vision Exercises on selective attention of the students. A 10-minutes of Bal-A-Vis-X training twice per week for eight weeks was administered. Significant gains in focused attention and concentration was reported and measured after the intervention in students.

A research investigating the effect of Bal-A-Vis-X protocol on elementary school students of special education department was carried on. A positive effect of Bal-A-Vis-X training is observed in on task attention during academic activities in children with ADHD , Autism and other mentally disabled individuals The past research records are evident that therapists have determined the individual effect of Aerobic training and Rhythmic Balance, Auditory, and Vision Exercises training for rehabilitation of ASD children. The evidence for implementation of two protocols for rehabilitation of ASD children is sparse. So the aim of this study is to compare the effects of Rhythmic Balance, Auditory, and Vision Exercises and Aerobic training in children with Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Give Consent to take part
* Children diagnosed with ASD by psychologist

Exclusion Criteria:

* Having co-morbidities like schizophrenia and developmental delay
* Showing aggressive behavior
* Having disease of cardiovascular or respiratory system
* Children with auditory and visual impairments

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Bruininks- Oseretsky Test of Motor Proficiency-2 (BOT-2) | 6 weeks
  Changes are measured from baseline. This test is used to measure 1. Fine Manual Control: Fine Motor Precision, Fine Motor Integration; 2. Manual Coordination: Manual Dexterity, Upper-Limb Coordination; 3. Body Coordination: Bilateral Coordination, Balance; 4. Strength and Agility: Running Speed and Agility.
Childhood Executive Functioning Inventory | 6 weeks
  Changes are measured from baseline. The Childhood Executive Functioning Inventory (CHEXI) is a rating instruments for parents and teachers that was developed in 2008 for measuring executive functioning in children.
Color Trail Test | 6 weeks
  Changes are measured from baseline. The Color Trails Test (CTT) is a language-free version of the Trail Making Test (TMT). The CTT is comprised of two tasks. The CTT manual reports that it takes 3-8 minutes to complete the CTT.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, MS-NMPT*, Principal Investigator — Riphah international university.pakistan
Locations (1):
- Child Dream Center, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No